CLINICAL TRIAL: NCT03932279
Title: Characterization of the Microbiome in Cutaneous T Cell Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Xiaolong (Alan) Zhou, Principal Investigator, Northwestern University
Other Study IDs: XZ05212018
Record Dates: First submitted 2019-02-18; First posted 2019-04-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Stage IA-IIA cutaneous T cell lymphoma
- Stage IIB and above cutaneous T cell lymphoma
- CD30+ lymphoproliferative disorders
- Plaque psoriasis with BSA>5% on routine phototherapy
- Moderate to severe atopic dermatitis on routine bleach bath
- Healthy controls

SUMMARY:
Investigators plan to perform a pilot study that aims to characterize the microbiome of human cutaneous T cell lymphoma patients and compare this to the microbiome of age and sex matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Patients with stage IA-IIA cutaneous T cell lymphoma
* Group 2: Patients with stage IIB and above cutaneous T cell lymphoma
* Group 3: Patients with CD30+ lymphoproliferative disorder including lymphomatoid papulosis and cutaneous anaplastic large cell lymphoma
* Group 4: Patients with plaque psoriasis with BSA>5% on routine phototherapy per standard of care
* Group 5: Patients with moderate to severe atopic dermatitis on routine bleach bath therapy per standard of care
* Group 6: Healthy individuals without the above skin conditions, similar age and sex distribution to the patients with cutaneous T cell lymphoma
* All Groups: subjects who are age 18-89 years of age at time of enrollment
* All Groups: Subjects who are able and willing to give informed consent for this study and the Dermatology Tissue Acquisition and Biorepository (STU00009443).

Exclusion Criteria:

* All Groups: Subjects who are younger than 18 years of age or older than 90 years of age
* All Groups: Subjects who are unable to give consent
* Patients currently on systemic antibiotics or recent (within past 4 weeks) exposure to systemic antibiotics
* We will not recruit the following populations: adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, prisoners and other vulnerable populations.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cutaneous T cell lymphoma, atopic dermatitis, and psoriasis and healthy individuals without any of these conditions will be enrolled at Northwestern Memorial Hospital Dermatology outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Bacterial diversity index | 3 months
  Diversity analysis of microbiome samples (measured by number of bacteria species/sample)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Zhou, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States